CLINICAL TRIAL: NCT02502344
Title: The Research About the Influence of Medical Interventions in the Period of Insulin Resistance on Prevalence of Abnormal Glucose Tolerance
Brief Title: Effect of Medical Interventions in Insulin Resistance on Prevalence of Abnormal Glucose Tolerance
Acronym: MIIIROPOAGT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12015C1023
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Insulin Resistance
Keywords: insulin resistance; abnormal glucose tolerance; DM prevention
MeSH Terms: conditions — Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- medical intervention group (Experimental): subjects in this group will accept healthy lifestyle changes such as food control and intensive exercise for 3 months first. Then their insulin resistance will be evaluated again . If their insulin resistance didn't improve, then they will take metformin 0.5g qd to reduce insulin resistance. If their insulin resistance improved, they will continued healthy lifestyle changes.
  Interventions: Behavioral: healthy lifestyle; Drug: Metformin
- clinical observeral group (No Intervention): subjects in this group will not accept medical interventions

INTERVENTIONS:
Behavioral: healthy lifestyle — food control and intensive exercise to lose weight
  Arms: medical intervention group
Drug: Metformin — use metformin to reduce insulin resistance
  Arms: medical intervention group

SUMMARY:
This research would take medical interventions in subjects of insulin resistance without abnormal glucose tolerance, to see if there were different prevalence of abnormal glucose tolerance in different groups.

DETAILED DESCRIPTION:
The situation of type 2 DM prevention in China is serious. The commonly accepted natural course of type 2 DM is as follows: obesity, insulin resistance(hyperinsulemia), abnormal glucose tolerance, DM and complications of DM; correspondently, the function status of pancreas islet β cells are: normal, compensatory, decompensatory, impaired and failure. Post researches have proved that using medical interventions after the period of insulin resistance when the function status of β cells were compensatory, the course could not be reversed. There were few clinical researches about effects of medical interventions in the period of insulin resistance . This research would take medical interventions in subjects of insulin resistance without abnormal glucose tolerance, to see if there were different prevalence of abnormal glucose tolerance in different groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 28kg/m2
* diagnosis of insulin resistance

Exclusion Criteria:

* abnormal glucose tolerance
* function impairment of heart, liver or kidney

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
prevalence of abnormal glucose intolerance | two years after the subject joins the research
  OGTT test will be took in these subjects to find out if their glucose tolerance was abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Jian Z Xiao, Doctor, Study Director — Beijing Tsinghua Changgeng Hospital
Locations (1):
- BEI JING Tsinghua Changguang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Ferrannini E, Mari A. beta-Cell function in type 2 diabetes. Metabolism. 2014 Oct;63(10):1217-27. doi: 10.1016/j.metabol.2014.05.012. Epub 2014 Jun 11. PMID 25070616
- [Background] Weir GC, Bonner-Weir S. Five stages of evolving beta-cell dysfunction during progression to diabetes. Diabetes. 2004 Dec;53 Suppl 3:S16-21. doi: 10.2337/diabetes.53.suppl_3.s16. PMID 15561905
- [Background] Samuel VT, Shulman GI. Mechanisms for insulin resistance: common threads and missing links. Cell. 2012 Mar 2;148(5):852-71. doi: 10.1016/j.cell.2012.02.017. PMID 22385956
- [Background] Li G, Zhang P, Wang J, Gregg EW, Yang W, Gong Q, Li H, Li H, Jiang Y, An Y, Shuai Y, Zhang B, Zhang J, Thompson TJ, Gerzoff RB, Roglic G, Hu Y, Bennett PH. The long-term effect of lifestyle interventions to prevent diabetes in the China Da Qing Diabetes Prevention Study: a 20-year follow-up study. Lancet. 2008 May 24;371(9626):1783-9. doi: 10.1016/S0140-6736(08)60766-7. PMID 18502303